CLINICAL TRIAL: NCT00644956
Title: A Randomized, Open-Label, Crossover, Multicenter, Single Dose Comparator Study Evaluating Onset Of Penile Rigidity In Men With Erectile Dysfunction Who Are Treated With Viagra (Sildenafil Citrate) And Cialis (Tadalafil)
Brief Title: A Randomized, Open-Label, Crossover, Multicenter, Single Dose Comparator Study Evaluating Onset Of Penile Rigidity In Men With Erectile Dysfunction Who Are Treated With Sildenafil And Tadalafil
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A1481183
Record Dates: First submitted 2008-03-25; First posted 2008-03-27 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — Tadalafil; Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Active Comparator)
  Interventions: Drug: sildenafil
- Arm 2 (Active Comparator)
  Interventions: Drug: tadalafil

INTERVENTIONS:
Drug: tadalafil — tadalafil 20 mg tablet by mouth for 2 doses (at Week 0 and Week 1)
  Arms: Arm 2
Drug: sildenafil — sildenafil 100 mg tablet by mouth for 2 doses (at Week 0 and Week 1)
  Arms: Arm 1

SUMMARY:
The objective of this study was to determine and compare the minimum time required to achieve penile rigidity greater than or equal to 60% at the base of the penis that is sustained for at least 3 minutes measured by Rigiscan®, following visual sexual stimulation post dose of 100 mg sildenafil citrate and 20 mg tadalafil in men with erectile dysfunction (ED).

ELIGIBILITY:
Inclusion Criteria:

* Included subjects were 18 years of age or older
* A clinical diagnosis of erectile dysfunction
* Known responders to either 100 mg sildenafil or 20 mg tadalafil.

Exclusion Criteria:

* Excluded were subjects who were unable to achieve penile rigidity of greater than or equal to 20% at the base of the penis that was sustained for at least 3 minutes
* Subjects who are able to achieve penile rigidity of greater than or equal to 60% at the base of the penis that was sustained for for at least 2 minutes or subjects who are able to achieve penile rigidity of greater than or equal to 80% at the base of the penis that is sustained for for at least 1 minute measured by Rigiscan®, at screening with no therapy, within 60 minutes following visual sexual stimulation
* Subjects currently using any commercially available treatments for erectile dysfunction
* Subjects on nitrates.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2003-06; Study Completion 2003-11 (Actual)

PRIMARY OUTCOMES:
The primary efficacy variable was time to onset of penile rigidity greater than or equal to 60% at the base of the penis, measured by Rigiscan, that was sustained for at least 3 minutes following visual sexual stimulation | Screening, Week 0, and Week 1

SECONDARY OUTCOMES:
The percentage of subjects who achieved penile rigidity greater than or equal to 60% at the base of the penis, measured by Rigiscan, that was sustained for at least 5 minutes following visual sexual stimulation | Screening, Week 0, and Week 1
Time to onset of penile rigidity greater than or equal to 60% at the base of the penis, measured by Regiscan, that was sustained for at least 5 minutes following visual sexual stimulation | Screening, Week 0, and Week 1
The percentage of subjects who achieved penile rigidity greater than or equal to 60% at the base of the penis, measured by Regiscan, that was sustained for at least 3 minutes following visual sexual stimulation | Screening, Week 0, and Week 1

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- Pfizer Investigational Site, Oslo, Norway
- Pfizer Investigational Site, Leeds, United Kingdom

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1481183&StudyName=A%20Randomized%2C%20Open-Label%2C%20Crossover%2C%20Multicenter%2C%20Single%20Dose%20Comparator%20Study%20Evaluating%20Onset%20Of%20Penile%20Rigidity%20In%20Men%20With%20Erect